CLINICAL TRIAL: NCT03705962
Title: Locally Applied Antibiotics for Infection Prophylaxis in Treatment of Open Fractures
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to continue study due to funding and personnel restraints
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Seth Yarboro, MD, Assistant Professor Orthopaedic Surgery, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18088
Record Dates: First submitted 2016-05-12; First posted 2018-10-15 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Fractures, Open
MeSH Terms: conditions — Fractures, Open | interventions — Tobramycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Antibiotic (Experimental): Subjects will be injected locally at the wound cavity (i.e. fracture site, surrounding soft tissue which include muscle, and subcutaneous space) with 80mg/40mL of tobramycin after wound closure. Systemic antibiotic will not be withheld and will be done along side the intervention.
  Interventions: Drug: Tobramycin
- Normal Saline (Placebo Comparator): Subjects will be injected locally with 40 mL 0.9% NS after wound closure. Systemic antibiotic will not be withheld and will be done along side the intervention.
  Interventions: Other: Placebo: normal saline

INTERVENTIONS:
Drug: Tobramycin
  Arms: Antibiotic
Other: Placebo: normal saline
  Arms: Normal Saline

SUMMARY:
The primary objective of this study is to investigate the effectiveness of local antibiotic versus placebo in the prevention of infections in open fractures. The study will assess whether local treatment of open fractures with the antibiotic tobramycin (in addition to standard systemic antibiotics) will decrease the risk and rate of infection, and rate of re-operation. This will be studied using a randomized controlled clinical trial design in adult population of age 18-70 years who present with open fractures. About 133 subjects will be recruited in this study at UVA.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 70 years
* Gustilo Type I,II,IIIa open fracture (s)
* Ability to provide informed consent (or proxy consent in cases where subject is temporarily impaired when intubated and sedated)
* Subject should be able to follow up at the scheduled times following surgery
* Subjects who may have compartment syndrome, renal insufficiency, and those who are immunosuppressed regardless of antibiotic administration will also be included in the study

Exclusion Criteria:

* Closed fracture
* Severe injury requiring flap coverage or vascular reconstruction (Gustilo-Anderson Type IIIB and C respectively)
* Aminoglycoside allergy
* Presentation greater than 48 hours after injury
* Pathologic fracture
* Preexisting infection in bone with an open fracture
* Patients with multiple trauma involving liver, kidney, or brain
* Pregnancy (self-reported)
* Current status as prisoner

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Yarboro, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Medical Center, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Antibiotic: Subjects will be injected locally at the wound cavity (i.e. fracture site, surrounding soft tissue which include muscle, and subcutaneous space) with 80mg/40mL of tobramycin after wound closure. Systemic antibiotic will not be withheld and will be done along side the intervention.
  Tobramycin
- Normal Saline: Subjects will be injected locally with 40 mL 0.9% NS after wound closure. Systemic antibiotic will not be withheld and will be done along side the intervention.
  Placebo: normal saline
Period: Overall Study
Arm/Group | Antibiotic | Normal Saline
Started | 8 | 3
Completed | 8 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects approached and enrolled presented to our emergency department with open fractures
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibiotic | Normal Saline | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 3 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Presence of Wound Infection
Description: Infection will be defined as major and minor, with major indicated by return to the operating room for irrigation and debridement. Minor infection is represented by documentation of cellulitis or superficial infection at surgical site and administration of oral antibiotics
Time Frame: 6 weeks post op
Population: We were only able to enroll 11 patients in this study. Our target n for recruitment for statistical significance was 120. Therefore, we did not perform statistical tests.
Measure: Count of Participants; unit: Participants
Arm/Group | Antibiotic | Normal Saline
Number analyzed (Participants) | 8 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks.
Arm/Group | Antibiotic | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/3
Other Adverse Events (participants affected / at risk) | 0/8 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antibiotic (N=8) | Normal Saline (N=3)
Suicide Ideation (Psychiatric disorders) | NA | 1

LIMITATIONS AND CAVEATS:
We were not able to enroll our goal of 120 patients; therefore, there is an insufficient sample size to perform any statistical test to evaluate the effect of early tobramycin in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT03705962/Prot_SAP_001.pdf
  • Informed Consent Form (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT03705962/ICF_000.pdf